CLINICAL TRIAL: NCT02706717
Title: Safety, Tolerability, and Effects of the Probiotic Visbiome Extra Strength on Gut Microbiome and Immune Activation Markers in HIV-Infected Participants on Suppressive Antiretroviral Therapy: A Phase II Study
Brief Title: Effects of the Probiotic Visbiome Extra Strength on Gut Microbiome & Immune Activation Markers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Exegi Pharma, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACTG A5350; 1U01AI068636 (NIH)
Record Dates: First submitted 2016-03-08; First posted 2016-03-11 (Estimated); Results first posted 2018-06-27 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2019-12

CONDITIONS: HIV-1 Infection

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Visbiome Extra Strength (Active Comparator)
  Interventions: Drug: Visbiome Extra Strength
- Placebo for Visbiome Extra Strength (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Visbiome Extra Strength — From week 2 to 4, participant will receive one sachet orally daily. From week 4 to 26, participant will receive one sachet orally twice daily.
  Arms: Visbiome Extra Strength
Drug: Placebo — From week 2 to 4, participant will receive one sachet orally daily. From week 4 to 26, participant will receive one sachet orally twice daily.
  Other Names: Control
  Arms: Placebo for Visbiome Extra Strength

SUMMARY:
The purpose of the study was to evaluate whether the probiotic Visbiome Extra Strength reduces inflammation in HIV-infected men and women when compared to a placebo (inactive medication like a dummy pill). The study evaluated whether taking Visbiome Extra Strength by mouth for 24 weeks was safe and well-tolerated for HIV-infected persons on antiretroviral therapy (ART). Probiotics are germs such as yeast or bacteria that are found in food and supplements that are used to improve the health of the digestive system. Many people refer to probiotics as "helpful bacteria." These bacteria live in the body and help the body work normally. In some medical conditions, including HIV infection, helpful bacteria are replaced with bacteria that can change the normal intestinal function and increase inflammation. The investigators tested whether giving a probiotic restored normal intestinal function and decreased inflammation.

DETAILED DESCRIPTION:
This was a phase II, randomized, double-blind, two-arm study to evaluate whether there is a significant change in sCD14 after 24 weeks of probiotic Visbiome Extra Strength (ES) therapy, and to determine the safety and tolerability of this agent in HIV-infected participants on stable antiretroviral therapy (ART). Participants were randomized 1:1 to Visbiome ES and placebo arms. Both arms initiated study treatment at Week 2 and took 1 sachet per day for the first 2 weeks and then 1 sachet twice daily for the next 22 weeks. All participants were followed for an additional 12 weeks off study product.

The study clinic visits included Entry (Week 0), and Weeks 2, 6, 14, 25, 26, and 38. Plasma for the primary outcome was collected at Weeks 0, 2, 25, and 26. The evaluations of safety (clinical assessment for signs and symptoms, diagnoses, and laboratory tests) were done at Weeks 2, 6, 14, 26, and 38.

Currently, the results are entered for the primary outcome measure and select secondary outcomes only. The results on the remaining secondary outcomes will be posted when they become available.

ELIGIBILITY:
Inclusion Criteria:

- HIV-1 infection, documented by any licensed rapid HIV test or HIV enzyme or chemiluminescence immunoassay (E/CIA) test kit at any time prior to study entry and confirmed by a licensed Western blot or a second antibody test by a method other than the initial rapid HIV and/or E/CIA, or by HIV-1 antigen, plasma HIV-1 RNA viral load.

NOTE: The term "licensed" refers to a US FDA-approved kit.

WHO (World Health Organization) and CDC (Centers for Disease Control and Prevention) guidelines mandate that confirmation of the initial test result must use a test that is different from the one used for the initial assessment. A reactive initial rapid test should be confirmed by either another type of rapid assay or an E/CIA that is based on a different antigen preparation and/or different test principle (eg, indirect versus competitive), or a Western blot or a plasma HIV-1 RNA viral load.

- Currently on continuous antiretroviral therapy (ART) for ≥48 weeks prior to study entry with no change in the ART regimen within the 24 weeks prior to study entry except as noted below.

NOTE A: Continuous ART is defined as continuous ART for the 48-week period prior to study entry with no ART interruption longer than 7 consecutive days.

NOTE B: Modifications of ART during the 24 weeks prior to study entry are permitted in certain circumstances. For example, the change in formulation (eg, from standard formulation to fixed-dose combination including ART modifications switching from ritonavir- to cobicistat-boosted protease inhibitors or from tenofovir disoproxil fumarate to tenofovir alafenamide) is allowed within 24 weeks prior to study entry. A within-class, single-drug substitution (eg, switch from nevirapine to efavirenz or from atazanavir to darunavir) is allowed within 24 weeks prior to study entry, with the exception of a switch between any other NRTI to/from abacavir. No other changes in ART within the 24 weeks prior to study entry are permitted.

* No plan to change ART regimen for the study duration.
* Screening CD4+ cell count >200 cells/mm3 obtained within 45 days prior to study entry by any US laboratory that has a CLIA certification or its equivalent.
* Screening HIV-1 RNA levels <50 copies/mL using a FDA-approved assay performed by any laboratory that has a CLIA certification or its equivalent within 45 days prior to study entry.
* HIV-1 RNA levels below the limit of quantification using a FDA-approved assay with a quantification limit of 50 copies/mL or lower for at least 48 weeks prior to study entry performed by any laboratory that has a CLIA certification or its equivalent.

NOTE: Single determinations that are between the assay quantification limit and 500 copies/mL (ie, "blips") are allowed as long as the preceding and subsequent determinations are below the level of quantification. The screening value may serve as the subsequent undetectable value following a blip.

* The following laboratory values obtained within 45 days prior to entry by any US laboratory that has a CLIA certification or its equivalent:

  * Absolute neutrophil count (ANC) ≥1000/mm3
  * Hemoglobin ≥10.0 g/dL for men and 9.0 g/dL for women
  * Platelet count ≥50,000/mm3
  * Aspartate aminotransferase (AST) (SGOT) ≤5 x upper limit normal (ULN)
  * Alanine aminotransferase (ALT) (SGPT) ≤5 x ULN
  * Alkaline phosphatase ≤5 x upper limit normal ULN
  * Total bilirubin ≤2.5 x ULN (if on atazanavir ≤5 x ULN)
  * Calculated creatinine clearance (CrCl) >60 mL/min, as estimated by the Cockcroft-Gault equation.
* For females of reproductive potential, negative serum or urine pregnancy test within 45 days prior to entry by any US clinic or laboratory that has a CLIA certification or its equivalent, or is using a point-of-care (POC)/ CLIA-waived test, or at any network-approved non-US laboratory or clinic that operates in accordance with Good Clinical Laboratory Practices (GCLP) and participates in appropriate external quality assurance programs.
* If participating in sexual activity that could lead to pregnancy, the female study participant must be willing to use a contraceptive while receiving protocol-specified medication. At least one of the following methods MUST be used:

  * Condoms (male or female), with or without a spermicidal agent
  * Diaphragm or cervical cap with spermicide
  * Intrauterine device (IUD)
  * Hormone-based contraceptive
* Ability and willingness of participant or legal guardian/representative to provide informed consent.

Exclusion Criteria:

- Initiation of ART during acute HIV infection.

NOTE: Participants who initiate ART within 6 months of HIV seroconversion are considered to have been initiated during acute infection and are excluded.

- Receipt of antibiotic therapy within 60 days prior to study entry.

NOTE: Antibiotics for opportunistic infection prophylaxis are exclusionary.

* Known allergy/sensitivity or any hypersensitivity to components of Visbiome Extra Strength or its formulation.
* Use of investigational therapies or investigational vaccines within 90 days prior to study entry.
* Non-investigational vaccinations within 2 weeks prior to study entry.
* Active drug or alcohol use or dependence that in the opinion of the site investigator would interfere with adherence to study requirements.
* Serious illness requiring systemic treatment and/or hospitalization within 30 days prior to entry.
* History of positive HCV antibody with detectable HCV RNA in plasma within 48 weeks prior to study entry.

NOTE: Persons with positive HCV Ab but negative plasma HCV RNA are allowed to participate. Sites must document negative HCV RNA within 24 weeks of study entry.

* History of positive HBsAg within 48 weeks prior to study entry.
* Liver cirrhosis, history of inflammatory bowel disease, total colectomy, colon or rectal anastomosis, bowel resection, or current colostomy.
* Current diagnosis of diabetes.
* Either breastfeeding or pregnant within 24 weeks prior to study entry.
* OIs within 45 days prior to study entry.
* Use of any of the following medications/products for more than 3 consecutive days within the 60 days prior to study entry:

  * Immunosuppressives (eg, azathioprine, corticosteroids greater than 20 mg per day [physiologic replacement doses are allowed], cyclosporine, mycophenolate, intravenous immunoglobulin (IVIG), interferon, sirolimus, sulfasalazine, tacrolimus).
  * Immune modulators (eg, cytokines [eg, IL-2], granulocyte colony stimulating factor, growth hormone, tumor necrosis factor antagonists, thalidomide).
  * Antineoplastic agents (except for topical agents for skin cancer).
  * Probiotics and prebiotics (supplements and products).

NOTE: Yogurt with live cultures is allowed.

* History of lactose intolerance or milk allergy.
* Any episode of acute or persistent diarrhea within 60 days prior to study entry.

NOTES:

1. Diarrhea is defined as three or more stools per day that are liquid/loose/watery and will take the shape of a container. If the duration of loose stools meeting this criterion definition is greater than 30 days, this is chronic diarrhea and is not exclusionary.
2. Acute diarrhea is defined as 3-14 day duration.
3. Persistent diarrhea is defined as 15-30 day duration.

   * Weight loss or gain of more than 25 pounds in the 24 weeks prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-06-05 (Actual); Study Completion 2017-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Andrade, MD, MPH, Study Chair — Johns Hopkins University; Edgar T Overton, MD, Study Chair — University of Alabama at Birmingham
Locations (25):
- United States (24):
  - 31788 Alabama CRS, Birmingham, Alabama
  - UCLA CARE Center CRS (601), Los Angeles, California
  - 701 University of California, San Diego AntiViral Research Center CRS, San Diego, California
  - 801 University of California, San Francisco HIV/AIDS CRS, San Francisco, California
  - University of Colorado Hospital CRS (6101), Aurora, Colorado
  - Northwestern University CRS (2701), Chicago, Illinois
  - Rush University Medical Center (2702), Chicago, Illinois
  - Johns Hopkins Adult AIDS CRS (201), Baltimore, Maryland
  - Washington University CRS (2101), St Louis, Missouri
  - 31786 New Jersey Medical School Clinical Research Center CRS, Newark, New Jersey
  - 7804 Weill Cornell Chelsea CRS, New York, New York
  - Columbia Physicians and Surgeons CRS (30329), New York, New York
  - 7803 Weill Cornell Upton CRS, New York, New York
  - Unc Aids Crs (3201), Chapel Hill, North Carolina
  - Greensboro CRS (3203), Greensboro, North Carolina
  - University of Cincinnati CRS (2401), Cincinnati, Ohio
  - Case CRS (2501), Cleveland, Ohio
  - The Ohio State University AIDS CRS (2301), Columbus, Ohio
  - 6201 Penn Therapeutics CRS, Philadelphia, Pennsylvania
  - Pittsburgh CRS (1001), Pittsburgh, Pennsylvania
  - Vanderbilt Therapeutics CRS (3652), Nashville, Tennessee
  - Trinity Health and Wellness Center CRS (31443), Dallas, Texas
  - Houston AIDS Research Team CRS (31473), Houston, Texas
  - University of Washington AIDS CRS (1401), Seattle, Washington
- Puerto Rico-AIDS CRS (5401), San Juan, Puerto Rico

REFERENCES:
- [Background] Chao, Anne. Scandinavian Journal of Statistics, 1 January 1984, Vol.11(4), pp.265-270
- [Background] Lemos LN, Fulthorpe RR, Triplett EW, Roesch LF. Rethinking microbial diversity analysis in the high throughput sequencing era. J Microbiol Methods. 2011 Jul;86(1):42-51. doi: 10.1016/j.mimet.2011.03.014. Epub 2011 Mar 30. PMID 21457733
- [Background] Magurran A. 2004. Measuring Biological Diversity. Blackwell Science Ltd, Oxford, United Kingdom
- See also: The Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Version 1.0, December 2004 (Clarification, August 2009). — https://rsc.tech-res.com/clinical-research-sites/safety-reporting/daids-grading-tables

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment began in 04/2016 and completed in 12/2016.
Groups:
- Visbiome Extra Strength: Visibiome: From week 2 to 4, participant will receive one sachet orally daily. From week 4 to 26, participant will receive one sachet orally twice daily.
Period: Overall Study
Arm/Group | Visbiome Extra Strength | Placebo for Visbiome Extra Strength
Started | 47 | 46 (3 placebo participants never initiated study treatment.)
Completed | 46 | 35
Not Completed | 1 | 11
Not completed — Withdrawal by Subject | 1 | 8
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Visbiome Extra Strength | Placebo for Visbiome Extra Strength | Total
Number analyzed (Participants) | 47 | 46 | 93
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 51 [47 to 56] | 51.5 [42 to 56] | 51 [45 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 40 | 40 | 80
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 9 | 19
  Not Hispanic or Latino | 37 | 37 | 74
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 21 | 17 | 38
  White | 24 | 26 | 50
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Puerto Rico | 1 | 0 | 1
  United States | 46 | 46 | 92
Smoking Status [Count of Participants; unit: Participants]
  Never | 15 | 19 | 34
  Former | 23 | 15 | 38
  Current | 9 | 10 | 19
  Unknown or Not Reported | 0 | 2 | 2
Alcohol Status [Count of Participants; unit: Participants]
  Never | 3 | 5 | 8
  Former | 15 | 8 | 23
  Current | 29 | 31 | 60
  Unknown or Not Reported | 0 | 2 | 2
Weight [Median (Inter-Quartile Range); unit: kg] | 87 [75.3 to 96.6] | 81.3 [71.7 to 94.1] | 83.1 [74.2 to 94.1]
BMI [Median (Inter-Quartile Range); unit: kg/m^2] — Population: One participant in the placebo arm did not have height collected on study and is thus missing BMI.
  kg/m^2
    number analyzed (Participants) | 47 | 45 | 92
    (all) | 27.3 [25.1 to 31.0] | 26.2 [23.6 to 30.1] | 27.1 [24.2 to 30.7]
CD4 Count [Median (Inter-Quartile Range); unit: cells/mm^3] | 702 [483 to 866] | 714.5 [546 to 897] | 712 [542 to 893]
HIV-1 RNA [Count of Participants; unit: Participants]
  <40 copies/mL | 47 | 45 | 92
  >=40 copies/mL | 0 | 1 | 1
sCD14 [Median (Inter-Quartile Range); unit: ug/L] | 2249 [2106 to 2759] | 2262 [2033 to 2643] | 2255 [2036 to 2750]

OUTCOME MEASURES:

1. Primary Outcome: Change in sCD14 From Baseline to Week 25/26
Description: Baseline is defined as the average of the Entry and Week 2 values. Week 25/26 is defined as the average of the Week 25 and Week 26 values.
  Absolute change was calculated as the value at Week 25/26 minus the value at Baseline.
Time Frame: Weeks 0, 2, 25, and 26
Population: Analysis used the per-protocol population. Participants 1) without Baseline AND Week 25/26 sCD14 values, or 2) with premature discontinuation of study treatment, or 3) or with HIV-1 virologic failure were excluded.
Measure: Mean (95% Confidence Interval); unit: ug/L
Arm/Group | Visbiome Extra Strength | Placebo for Visbiome Extra Strength
Number analyzed (Participants) | 42 | 31
ug/L | 41 [-94.1 to 176.2] | 92.3 [-48.5 to 233.2]
Statistical Analysis 1: Comparison: Visbiome Extra Strength vs Placebo for Visbiome Extra Strength; Test type: Superiority; p = 0.60, t-test, 2 sided; 2-sample t-test with equal variance; Mean Difference (Net) = -51.3, 95% CI 2-sided [-246 to 143.9] — Mean difference is Visbiome ES mean minus placebo mean

2. Secondary Outcome: Change in IL-6 From Week 2 to Week 26
Description: IL-6 data are not available as of June, 2018. These data are based on assays which are to be tested in batch to minimize variability. Due to batch testing, shipment of samples for testing could not begin until after the study follow-up completion, which was 3 months after the primary completion date. Please note that these secondary outcomes were not included in the primary analysis report. There are many outcomes in this study and the labs had to give priority to the assays planned to be included in the primary manuscript.
Time Frame: Weeks 2 and 26
Population: These data were not assayed and the analysis was abandoned.
Arm/Group | Visbiome Extra Strength | Placebo for Visbiome Extra Strength
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change in IP-10 From Week 2 to Week 26
Description: All values were log10 transformed prior to calculating change and conducting analyses.
  Absolute change was calculated as the value at Week 26 minus the value at Week 2. Mean changes were exponentiated to be back on the untransformed scale and corresponds to a mean fold change.
Time Frame: Weeks 2 and 26
Population: Analysis used the per-protocol population. Participants 1) without Baseline AND Week 25/26 sCD14 values, or 2) with premature discontinuation of study treatment, or 3) or with HIV-1 virologic failure were excluded. Additionally, participants without Week 2 and Week 26 IP-10 data were excluded.
Measure: Mean (95% Confidence Interval); unit: Fold change
Arm/Group | Visbiome Extra Strength | Placebo for Visbiome Extra Strength
Number analyzed (Participants) | 42 | 30
Fold change | 1.05 [0.80 to 1.38] | 0.94 [0.75 to 1.18]

4. Secondary Outcome: Change in sCD163 From Week 2 to Week 26
Description: sCD163 data are not available as of June, 2018. These data are based on assays which are to be tested in batch to minimize variability. Due to batch testing, shipment of samples for testing could not begin until after the study follow-up completion, which was 3 months after the primary completion date. Please note that these secondary outcomes were not included in the primary analysis report. There are many outcomes in this study and the labs had to give priority to the assays planned to be included in the primary manuscript.
Time Frame: Weeks 2 and 26
Population: These data were not assayed and the analysis was abandoned.
Arm/Group | Visbiome Extra Strength | Placebo for Visbiome Extra Strength
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in sTNF-RI From Week 2 to Week 26
Description: sTNF-RI data are not available as of June, 2018. These data are based on assays which are to be tested in batch to minimize variability. Due to batch testing, shipment of samples for testing could not begin until after the study follow-up completion, which was 3 months after the primary completion date. Please note that these secondary outcomes were not included in the primary analysis report. There are many outcomes in this study and the labs had to give priority to the assays planned to be included in the primary manuscript.
Time Frame: Weeks 2 and 26
Population: These data were not assayed and the analysis was abandoned.
Arm/Group | Visbiome Extra Strength | Placebo for Visbiome Extra Strength
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change in Oxidized LDL From Week 2 to Week 26
Description: Oxidized LDL data are not available as of June, 2018. These data are based on assays which are to be tested in batch to minimize variability. Due to batch testing, shipment of samples for testing could not begin until after the study follow-up completion, which was 3 months after the primary completion date. Please note that these secondary outcomes were not included in the primary analysis report. There are many outcomes in this study and the labs had to give priority to the assays planned to be included in the primary manuscript.
Time Frame: Weeks 2 and 26
Population: These data were not assayed and the analysis was abandoned.
Arm/Group | Visbiome Extra Strength | Placebo for Visbiome Extra Strength
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change in Kynurenine to Tryptophan Ratio From Week 2 to Week 26
Description: Fold change was calculated as the value at Week 26 divided by the value at Week 2.
Time Frame: Weeks 2 and 26
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | Visbiome Extra Strength | Placebo for Visbiome Extra Strength
Number analyzed (Participants) | 42 | 31
ratio | 1.039 [0.935 to 1.143] | 0.997 [0.944 to 1.05]
Statistical Analysis 1: Comparison: Visbiome Extra Strength vs Placebo for Visbiome Extra Strength; Test type: Superiority; p = 0.51, t-test, 2 sided; 2-sample t-test with equal variance; Mean Difference (Net) = 0.042, 95% CI 2-sided [-0.09 to 0.17] — Mean difference is Visbiome ES mean minus placebo mean

8. Secondary Outcome: Change in D-dimer From Week 2 to Week 26
Description: as for outcome 3
Time Frame: Weeks 2 and 26
Population: Analysis used the per-protocol population. Participants 1) without Baseline AND Week 25/26 sCD14 values, or 2) with premature discontinuation of study treatment, or 3) or with HIV-1 virologic failure were excluded. Additionally, participants without Week 2 and Week 26 D-dimer data were excluded.
Measure: Mean (95% Confidence Interval); unit: Fold change
Arm/Group | Visbiome Extra Strength | Placebo for Visbiome Extra Strength
Number analyzed (Participants) | 40 | 31
Fold change | 1.203 [0.967 to 1.496] | 0.937 [0.787 to 1.115]
Statistical Analysis 1: Comparison: Visbiome Extra Strength vs Placebo for Visbiome Extra Strength; Test type: Superiority; p = 0.09, t-test, 2 sided; 2-sample t-test with equal variance; Mean Difference (Net) = 28.4, 95% CI 2-sided [-3.6 to 71.0] — The estimation parameter is the percent difference between the geometric mean fold changes. With d-dimer data log10 transformed, this is (exp(Visbiome ES mean minus placebo mean) - 1)*100

9. Secondary Outcome: Change in LPS From Week 2 to Week 26
Description: LPS data are not available as of June, 2018. These data are based on assays which are to be tested in batch to minimize variability. Due to batch testing, shipment of samples for testing could not begin until after the study follow-up completion, which was 3 months after the primary completion date. Please note that these secondary outcomes were not included in the primary analysis report. There are many outcomes in this study and the labs had to give priority to the assays planned to be included in the primary manuscript.
Time Frame: Weeks 2 and 26
Population: These data were not assayed and the analysis was abandoned.
Arm/Group | Visbiome Extra Strength | Placebo for Visbiome Extra Strength
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Change in LBP From Week 2 to Week 26
Description: LBP data are not available as of June, 2018. These data are based on assays which are to be tested in batch to minimize variability. Due to batch testing, shipment of samples for testing could not begin until after the study follow-up completion, which was 3 months after the primary completion date. Please note that these secondary outcomes were not included in the primary analysis report. There are many outcomes in this study and the labs had to give priority to the assays planned to be included in the primary manuscript.
Time Frame: Weeks 2 and 26
Population: These data were not assayed and the analysis was abandoned.
Arm/Group | Visbiome Extra Strength | Placebo for Visbiome Extra Strength
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Change in CD4+ Cell Count From Week 2 to Week 26.
Description: Absolute change was calculated as the value at Week 26 minus the value at Week 2.
Time Frame: Weeks 2 and 26
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: cells/mm^3
Arm/Group | Visbiome Extra Strength | Placebo for Visbiome Extra Strength
Number analyzed (Participants) | 42 | 31
cells/mm^3 | 9.8 [-31.7 to 51.2] | 42.4 [-2.7 to 87.6]
Statistical Analysis 1: Comparison: Visbiome Extra Strength vs Placebo for Visbiome Extra Strength; Test type: Superiority; p = 0.29, t-test, 2 sided; 2-sample t-test with equal variance; Mean Difference (Net) = -32.7, 95% CI 2-sided [-93.5 to 28.2] — Mean difference is Visbiome ES mean minus placebo mean

12. Secondary Outcome: Change in CD4+/CD8+ Ratio From Week 2 to Week 26.
Description: Fold change was calculated as the value at Week 26 divided by the value at Week 2.
Time Frame: Weeks 2 and 26
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | Visbiome Extra Strength | Placebo for Visbiome Extra Strength
Number analyzed (Participants) | 42 | 31
ratio | 1.03 [0.99 to 1.07] | 1.05 [1.01 to 1.09]
Statistical Analysis 1: Comparison: Visbiome Extra Strength vs Placebo for Visbiome Extra Strength; Test type: Superiority; p = 0.41, t-test, 2 sided; 2-sample t-test with equal variance; Mean Difference (Net) = -0.02, 95% CI 2-sided [-0.08 to 0.04] — Mean difference is Visbiome ES mean minus placebo mean

13. Secondary Outcome: Change in %CD14++CD16- From Week 2 to Week 26.
Description: Absolute change was calculated as the value at Week 26 minus the value at Week 2.
Time Frame: Weeks 2 and 26
Population: Analysis used the per-protocol population. Participants 1) without Baseline AND Week 25/26 sCD14 values, or 2) with premature discontinuation of study treatment, or 3) or with HIV-1 virologic failure were excluded. Additionally, participants without Week 2 and Week 26 %CD14++CD16- data were excluded.
Measure: Mean (95% Confidence Interval); unit: Percent of %CD14++CD16- cells
Arm/Group | Visbiome Extra Strength | Placebo for Visbiome Extra Strength
Number analyzed (Participants) | 41 | 28
Percent of %CD14++CD16- cells | 2.18 [-1.16 to 5.53] | -1.25 [-3.31 to 0.80]

14. Secondary Outcome: Change in %CD14++CD16+ From Week 2 to Week 26
Description: Absolute change was calculated as the value at Week 26 minus the value at Week 2.
Time Frame: Weeks 2 and 26
Population: Analysis used the per-protocol population. Participants 1) without Baseline AND Week 25/26 sCD14 values, or 2) with premature discontinuation of study treatment, or 3) or with HIV-1 virologic failure were excluded. Additionally, participants without Week 2 and Week 26 %CD14++CD16+ data were excluded.
Measure: Mean (95% Confidence Interval); unit: Percent of %CD14++CD16+ cells
Arm/Group | Visbiome Extra Strength | Placebo for Visbiome Extra Strength
Number analyzed (Participants) | 41 | 28
Percent of %CD14++CD16+ cells | 0.81 [-0.02 to 1.64] | 0.47 [-0.19 to 1.12]

15. Secondary Outcome: Change in %CD14lowCD16hi From Week 2 to Week 26
Description: %CD14lowCD16hi data are not available as of June, 2018. These data are based on assays which are to be tested in batch to minimize variability. Due to batch testing, shipment of samples for testing could not begin until after the study follow-up completion, which was 3 months after the primary completion date. Please note that these secondary outcomes were not included in the primary analysis report. There are many outcomes in this study and the labs had to give priority to the assays planned to be included in the primary manuscript.
Time Frame: Weeks 2 and 26
Population: These data were not assayed and the analysis was abandoned.
Arm/Group | Visbiome Extra Strength | Placebo for Visbiome Extra Strength
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Change in %CD4+CD38+ From Week 2 to Week 26.
Description: %CD4+CD38+ data are not available as of June, 2018. These data are based on assays which are to be tested in batch to minimize variability. Due to batch testing, shipment of samples for testing could not begin until after the study follow-up completion, which was 3 months after the primary completion date. Please note that these secondary outcomes were not included in the primary analysis report. There are many outcomes in this study and the labs had to give priority to the assays planned to be included in the primary manuscript.
Time Frame: Weeks 2 and 26
Population: These data were not assayed and the analysis was abandoned.
Arm/Group | Visbiome Extra Strength | Placebo for Visbiome Extra Strength
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Change in %CD4+HLA-DR+ From Week 2 to Week 26.
Description: %CD4+HLA-DR+ data are not available as of June, 2018. These data are based on assays which are to be tested in batch to minimize variability. Due to batch testing, shipment of samples for testing could not begin until after the study follow-up completion, which was 3 months after the primary completion date. Please note that these secondary outcomes were not included in the primary analysis report. There are many outcomes in this study and the labs had to give priority to the assays planned to be included in the primary manuscript.
Time Frame: Weeks 2 and 26
Population: These data were not assayed and the analysis was abandoned.
Arm/Group | Visbiome Extra Strength | Placebo for Visbiome Extra Strength
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Change in %CD4+CD38+HLA-DR+ From Week 2 to Week 26.
Description: Absolute change was calculated as the value at Week 26 minus the value at Week 2.
Time Frame: Weeks 2 and 26
Population: Analysis used the per-protocol population. Participants 1) without Baseline AND Week 25/26 sCD14 values, or 2) with premature discontinuation of study treatment, or 3) or with HIV-1 virologic failure were excluded. Additionally, participants without Week 2 and Week 26 %CD4+CD38+HLA-DR+ data were excluded.
Measure: Mean (95% Confidence Interval); unit: Percent of %CD4+CD38+HLA-DR+ cells
Arm/Group | Visbiome Extra Strength | Placebo for Visbiome Extra Strength
Number analyzed (Participants) | 41 | 28
Percent of %CD4+CD38+HLA-DR+ cells | -0.06 [-0.25 to 0.29] | -0.07 [-0.28 to 0.14]

19. Secondary Outcome: Change in %CD8+CD38+ From Week 2 to Week 26.
Description: %CD8+CD38+ data are not available as of June, 2018. These data are based on assays which are to be tested in batch to minimize variability. Due to batch testing, shipment of samples for testing could not begin until after the study follow-up completion, which was 3 months after the primary completion date. Please note that these secondary outcomes were not included in the primary analysis report. There are many outcomes in this study and the labs had to give priority to the assays planned to be included in the primary manuscript.
Time Frame: Weeks 2 and 26
Population: These data were not assayed and the analysis was abandoned.
Arm/Group | Visbiome Extra Strength | Placebo for Visbiome Extra Strength
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Change in %CD8+HLA-DR+ From Week 2 to Week 26.
Description: %CD8+HLA-DR+ data are not available as of June, 2018. These data are based on assays which are to be tested in batch to minimize variability. Due to batch testing, shipment of samples for testing could not begin until after the study follow-up completion, which was 3 months after the primary completion date. Please note that these secondary outcomes were not included in the primary analysis report. There are many outcomes in this study and the labs had to give priority to the assays planned to be included in the primary manuscript.
Time Frame: Weeks 2 and 26
Population: These data were not assayed and the analysis was abandoned.
Arm/Group | Visbiome Extra Strength | Placebo for Visbiome Extra Strength
Number analyzed (Participants) | 0 | 0

21. Secondary Outcome: Change in %CD8+CD38+HLA-DR+ From Week 2 to Week 26.
Description: Absolute change was calculated as the value at Week 26 minus the value at Week 2.
Time Frame: Weeks 2 and 26
Population: Analysis used the per-protocol population. Participants 1) without Baseline AND Week 25/26 sCD14 values, or 2) with premature discontinuation of study treatment, or 3) or with HIV-1 virologic failure were excluded. Additionally, participants without Week 2 and Week 26 %CD8+CD38+HLA-DR+ data were excluded.
Measure: Mean (95% Confidence Interval); unit: Percent of %CD8+CD38+HLA-DR+ cells
Arm/Group | Visbiome Extra Strength | Placebo for Visbiome Extra Strength
Number analyzed (Participants) | 41 | 28
Percent of %CD8+CD38+HLA-DR+ cells | 0.19 [-0.47 to 0.86] | -0.13 [-0.78 to 0.53]

22. Secondary Outcome: Change in %CD4+CD28-CD57+ From Week 2 to Week 26.
Description: Absolute change was calculated as the value at Week 26 minus the value at Week 2.
Time Frame: Weeks 2 and 26
Population: Analysis used the per-protocol population. Participants 1) without Baseline AND Week 25/26 sCD14 values, or 2) with premature discontinuation of study treatment, or 3) or with HIV-1 virologic failure were excluded. Additionally, participants without Week 2 and Week 26 %CD4+CD28-CD57+ data were excluded.
Measure: Mean (95% Confidence Interval); unit: Percent of %CD4+CD28-CD57+ cells
Arm/Group | Visbiome Extra Strength | Placebo for Visbiome Extra Strength
Number analyzed (Participants) | 41 | 28
Percent of %CD4+CD28-CD57+ cells | -0.08 [-0.57 to 0.40] | -0.09 [-0.72 to 0.53]

23. Secondary Outcome: Change in %CD8+CD28-CD57+ From Week 2 to Week 26.
Description: Absolute change was calculated as the value at Week 26 minus the value at Week 2.
Time Frame: Weeks 2 and 26
Population: Analysis used the per-protocol population. Participants 1) without Baseline AND Week 25/26 sCD14 values, or 2) with premature discontinuation of study treatment, or 3) or with HIV-1 virologic failure were excluded. Additionally, participants without Week 2 and Week 26 %CD8+CD28-CD57+ data were excluded.
Measure: Mean (95% Confidence Interval); unit: Percent of %CD8+CD28-CD57+ cells
Arm/Group | Visbiome Extra Strength | Placebo for Visbiome Extra Strength
Number analyzed (Participants) | 41 | 28
Percent of %CD8+CD28-CD57+ cells | 0.77 [-0.59 to 2.13] | -1.50 [-3.36 to 0.35]

24. Secondary Outcome: Change in Chao1 Richness Index From Week 2 to Week 26.
Description: Absolute change was calculated as the value at Week 26 minus the value at Week 2.
  Chao1 is a diversity index that reflects how many different quantifiable types (species, individuals, items, etc…) there are in a dataset (see Chao reference). Chao1 diversity is a richness measure which quantifies how many different types there are in a given dataset. The Chao 1 index can range from 1 to infinity as it is constrained only by the number of types defined as measurable. The greater a value is, the more diverse it is but only in direct comparison to groups considering the same parameters. That is, diversity indices are relative to the community (cohort or ecosystem) studied in part due to the definition of the "types" that are considered.
Time Frame: Weeks 2 and 26
Population: Analysis used the per-protocol population. Participants 1) without Baseline AND Week 25/26 sCD14 values, or 2) with premature discontinuation of study treatment, or 3) or with HIV-1 virologic failure were excluded. Additionally, participants without Week 2 and Week 26 Chao1 richness index data were excluded.
Measure: Mean (95% Confidence Interval); unit: Estimator of species richness
Arm/Group | Visbiome Extra Strength | Placebo for Visbiome Extra Strength
Number analyzed (Participants) | 29 | 21
Estimator of species richness | 48.8 [-151 to 249] | 78.2 [-205 to 362]

25. Secondary Outcome: Change in Shannon Diversity Index From Week 2 to Week 26.
Description: Absolute change was calculated as the value at Week 26 minus the value at Week 2.
  Shannon is a diversity index that reflects how many different quantifiable types (species, individuals, items, etc…) there are in a dataset (see Lemos and Magurran references). The Shannon index is an estimator of richness and evenness. It quantifies uncertainty (entropy) within a dataset. The Shannon Index ranges from 0-5. The greater a value is, the more diverse it is but only in direct comparison to groups considering the same parameters. That is, diversity indices are relative to the community (cohort or ecosystem) studied in part due to the definition of the "types" that are considered.
Time Frame: Weeks 2 and 26
Population: Analysis used the per-protocol population. Participants 1) without Baseline AND Week 25/26 sCD14 values, or 2) with premature discontinuation of study treatment, or 3) or with HIV-1 virologic failure were excluded. Additionally, participants without Week 2 and Week 26 Shannon diversity index data were excluded.
Measure: Mean (95% Confidence Interval); unit: Estimator of species richness & evenness
Arm/Group | Visbiome Extra Strength | Placebo for Visbiome Extra Strength
Number analyzed (Participants) | 29 | 21
Estimator of species richness & evenness | 0.11 [-0.09 to 0.32] | 0.13 [-0.21 to 0.47]

26. Secondary Outcome: Change in Chao1 Richness Index From Week 26 to Week 38.
Description: Absolute change was calculated as the value at Week 38 minus the value at Week 26.
  Chao1 is a diversity index that reflects how many different quantifiable types (species, individuals, items, etc…) there are in a dataset (see Chao reference). Chao1 diversity is a richness measure which quantifies how many different types there are in a given dataset. The Chao 1 index can range from 1 to infinity as it is constrained only by the number of types defined as measurable. The greater a value is, the more diverse it is but only in direct comparison to groups considering the same parameters. That is, diversity indices are relative to the community (cohort or ecosystem) studied in part due to the definition of the "types" that are considered.
Time Frame: Weeks 26 and 38
Population: Analysis used the per-protocol population. Participants 1) without Baseline AND Week 25/26 sCD14 values, or 2) with premature discontinuation of study treatment, or 3) or with HIV-1 virologic failure were excluded. Additionally, participants without Week 26 and Week 38 Chao1 richness index data were excluded.
Measure: Mean (95% Confidence Interval); unit: Estimator of species richness
Arm/Group | Visbiome Extra Strength | Placebo for Visbiome Extra Strength
Number analyzed (Participants) | 29 | 22
Estimator of species richness | 23 [-227 to 273] | -14.1 [-385 to 357]

27. Secondary Outcome: Change in Shannon Diversity Index From Week 26 to Week 38.
Description: Absolute change was calculated as the value at Week 38 minus the value at Week 26.
  Shannon is a diversity index that reflects how many different quantifiable types (species, individuals, items, etc…) there are in a dataset (see Lemos and Magurran references). The Shannon index is an estimator of richness and evenness. It quantifies uncertainty (entropy) within a dataset. The Shannon Index ranges from 0-5. The greater a value is, the more diverse it is but only in direct comparison to groups considering the same parameters. That is, diversity indices are relative to the community (cohort or ecosystem) studied in part due to the definition of the "types" that are considered.
Time Frame: Weeks 26 and 38
Population: Analysis used the per-protocol population. Participants 1) without Baseline AND Week 25/26 sCD14 values, or 2) with premature discontinuation of study treatment, or 3) or with HIV-1 virologic failure were excluded. Additionally, participants without Week 26 and Week 38 Shannon diversity index data were excluded.
Measure: Mean (95% Confidence Interval); unit: Estimator of species richness & evenness
Arm/Group | Visbiome Extra Strength | Placebo for Visbiome Extra Strength
Number analyzed (Participants) | 29 | 22
Estimator of species richness & evenness | -0.10 [-0.46 to 0.26] | 0.03 [-0.35 to 0.41]

28. Secondary Outcome: Change in I-FABP From Week 2 to Week 26.
Description: Absolute change was calculated as the value at Week 26 minus the value at Week 2.
Time Frame: Weeks 2 and 26
Population: Analysis used the per-protocol population. Participants 1) without Baseline AND Week 25/26 sCD14 values, or 2) with premature discontinuation of study treatment, or 3) or with HIV-1 virologic failure were excluded. Additionally, participants without Week 2 and Week 26 I-FABP data were excluded.
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Visbiome Extra Strength | Placebo for Visbiome Extra Strength
Number analyzed (Participants) | 42 | 30
ng/mL | 0.59 [0.26 to 1.34] | 0.83 [0.37 to 1.86]

29. Secondary Outcome: Safety
Description: Summary of the highest adverse event grade (0-5) for each participant.
  Protocol definition of Adverse Events: 1) signs and symptoms Grade ≥3 and any that led to a change in treatment regardless of grade; 2) new diagnoses; 3) Grade ≥3 lab values and any that led to a change in treatment or were associated with a diagnosis were recorded, regardless of grade.
  DAIDS AE Grading Table, Version 2.0 was used.
Time Frame: Treatment dispensation to Week 38
Population: All enrolled participants who initiated study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Visbiome Extra Strength | Placebo for Visbiome Extra Strength
Number analyzed (Participants) | 47 | 43
Participants
  Grade 0 | 32 | 35
  Grade 1 | 3 | 3
  Grade 2 | 5 | 1
  Grade 3 | 5 | 3
  Grade 4 | 2 | 0
  Grade 5 | 0 | 1
Statistical Analysis 1: Comparison: Visbiome Extra Strength vs Placebo for Visbiome Extra Strength; Test type: Superiority; p = 0.15, Kruskal-Wallis

30. Secondary Outcome: Tolerability
Description: Tolerability was successfully completing the protocol-defined treatment period.
Time Frame: Treatment dispensation to Week 38
Population: All enrolled participants who initiated study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Visbiome Extra Strength | Placebo for Visbiome Extra Strength
Number analyzed (Participants) | 47 | 43
Participants
  Completed as defined by protocol | 43 | 31
  Did not complete as defined by protocol | 4 | 12

ADVERSE EVENTS:
Time Frame: Week 0 to Week 38.
Description: Protocol definition of Adverse Events: 1) signs and symptoms Grade ≥3 and any that led to a change in treatment regardless of grade; 2) new diagnoses; 3) Grade ≥3 lab values and any that led to a change in treatment or were associated with a diagnosis were recorded, regardless of grade.
  DAIDS AE Grading Table, Version 2.0 was used.
Arm/Group | Visbiome Extra Strength | Placebo for Visbiome Extra Strength
All-Cause Mortality (participants affected / at risk) | 0/47 | 1/46
Serious Adverse Events (participants affected / at risk) | 5/47 | 2/46
Other Adverse Events (participants affected / at risk) | 0/47 | 0/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Visbiome Extra Strength (N=47) | Placebo for Visbiome Extra Strength (N=46)
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Meningoencephalitis herpetic (Infections and infestations) | 0 | 1
Comminuted fracture (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2016-04-15): https://cdn.clinicaltrials.gov/large-docs/17/NCT02706717/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-06): https://cdn.clinicaltrials.gov/large-docs/17/NCT02706717/SAP_001.pdf